CLINICAL TRIAL: NCT07296783
Title: Transforming Research and Clinical Knowledge in Geriatric Traumatic Brain Injury (TRACK-GERI)
Acronym: TRACK-GERI
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Doris Duke Charitable Foundation (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute on Aging (NIA) (NIH); United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: TRACK-GERI; 1R01NS110944 (NIH); K23NS095755 (NIH); 1K76AG083285 (NIH); W81XWH2110469 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2025-12-16; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will undergo phlebotomy for whole blood collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- TRACK-GERI TBI Patients: TBI patients
- TRACK-GERI Study Partners of TBI Patients: Study partners of TBI patients
- TRACK-GERI Controls: Controls
- TRQACK-GERI Study Partners of Control Patients: Study partners of control patients
- TRACK-VA TBI Patients: VA TBI patients
- TRACK-VA Study Partners of TBI Patients: Study partners of VA TBI patients
- TRACK-VA Controls: VA controls
- TRACK-VA Study Partners of Control Patients: Study partners of VA control patients

SUMMARY:
The purpose of this study is to improve the diagnosis and prediction of recovery after traumatic brain injury (TBI) in adults age 65 years and older. The study will follow older adults who present to the emergency department after TBI, as well as matched control participants, and will measure clinical features, brain imaging, and blood-based biomarkers over 12 months to understand how recovery changes over time. Researchers will examine how pre-injury health, brain structure, and biological markers are related to disability and cognitive outcomes after TBI. Information from this study will be used to develop age-appropriate tools to better diagnose TBI and estimate long-term outcomes in older adults.

ELIGIBILITY:
TRACK-GERI/VA TBI PATIENT INCLUSION/EXCLUSION CRITERIA

Inclusion Criteria:

1. Age 65 years and older, no upper age limit
2. Reliable report or physical evidence of head trauma
3. Injury occurred <72 hours ago (within 14 days of injury for TRACK-VA TBI patients)
4. Acute brain CT for clinical use
5. Fluency in English/Chinese (UCSF only)
6. Ability to obtain informed consent from subject or legally authorized representative
7. Ability to be co-enrolled with a study partner who meets Study Partner enrollment criteria

Exclusion Criteria:

1. Significant polytrauma that would interfere with follow-up and outcome assessment
2. Prisoners or patients in custody
3. Patients on psychiatric hold (e.g. 5150, 5250)
4. Low likelihood follow-up (participant or family is indicating a low interest, homelessness, out of state/country)
5. Current participation in an interventional trial
6. Penetrating TBI
7. Spinal cord injury with ASIA score of C or worse
8. Acute disabling neurological injury (e.g. acute stroke, cardiac arrest concurrent with head trauma presentation)

TRACK-GERI/VA STUDY PARTNERS OF TBI PATIENTS INCLUSION/EXCLUSION CRITERIA

Inclusion Criteria:

1. Age 18 years or older
2. Either designated by the patient, presents with patient to the Emergency Department, is listed in the patient's medical chart as an alternate/emergency contact, or is the patient's case manager/social worker, and knows the patient well enough to comment on the patient's health and functional status (e.g. may be family member, friend, caregiver, case manager, etc).
3. Ability to read, write, and speak English/Chinese (UCSF only)
4. Ability to provide informed consent for self

Exclusion Criteria:

1. Pre-existing and major disabling medical, psychiatric, or other neurological disease (e.g. dementia) that interferes with ability to provide evaluation of patient's health and functional status.
2. Prisoners or patients in custody
3. Patients on psychiatric hold (e.g. 5150, 5250)

TRACK-GERI/VA CONTROL SUBJECT INCLUSION/EXCLUSION CRITERIA

Inclusion Criteria:

1. Age 65 years or older, no upper age limit
2. Visual acuity/hearing adequate for testing
3. Fluency in English/Chinese (UCSF only)
4. Ability to obtain informed consent from subject or legally authorized representative
5. Ability to be co-enrolled with a study partner who meets study partner enrollment criteria (see control study partner enrollment criteria)
6. For TRACK-VA patients only: Presentation to SFVAMC ED for acute care with planned discharge from ED.

Exclusion Criteria:

1. Medically diagnosed with traumatic brain or orthopedic injury in the last year (TRACK-VA Control Subjects are not excluded for orthopedic injuries)
2. Significant polytrauma that would interfere with follow-up and outcome assessment
3. Prisoners or patients in custody
4. Patients on psychiatric hold (e.g. 5150, 5250)
5. Low likelihood follow-up (participant or family is indicating low interest, homelessness, out of state/country)
6. Current participation in an interventional trial
7. Penetrating TBI
8. Spinal cord injury with ASIA score of C or worse
9. Acute disabling neurological injury (e.g. acute stroke, cardiac arrest)

TRACK-GERI/VA STUDY PARTNERS OF CONTROL SUBJECTS INCLUSION/EXCLUSION CRITERIA

Inclusion Criteria:

1. Age 18 years or older
2. Designated by the control subject as someone who knows the subject well enough to comment on their health and functional starus (e.g., may be family member, friend, caregiver, case manager, etc.)
3. Ability to read, write and speak English/Chinese (UCSF only)
4. Ability to provide informed consent for self

Exclusion Criteria:

1. Pre-existing and major disabling medical, psychiatric, or other neurological disease (e.g. dementia) that interferes with ability to provide evaluation of control subject's health and functional status.
2. Prisoners or in custody
3. On psychiatric hold (e.g. 5150, 5250)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants are those with and without TBI, along with study partners.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome at 6 Months Post-Injury as Assessed by the Glasgow Outcome Scale-Extended (GOSE) | 6 months post-injury
  Functional outcome after traumatic brain injury will be measured using the Glasgow Outcome Scale-Extended (GOSE). The score ranges from 1-8, with higher scores indicating better recovery. The primary outcome is GOSE assessed at 6 months post-injury.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Manley, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through the Federal Interagency TBI Research (FITBIR) Database.
Time Frame: Shared scientific data will be made accessible as soon as possible, and no later than the time of an associated publication, or the end of performance period, whichever comes first.
Access Criteria: FITBIR qualified investigators will be provided access.
URL: https://fitbir.nih.gov/

REFERENCES:
- See also: Related Info — https://tracktbi.ucsf.edu/
- See also: Related Info — https://tracktbi.ucsf.edu/publications
- See also: Related Info — https://tracktbinet.ucsf.edu/